CLINICAL TRIAL: NCT05532098
Title: Comparative Efficacy of Platelet Rich Plasma and Dry Needling in Management of Anterior Disc Displacement of Temporomandibular Joint
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SURIYA N OMR
Record Dates: First submitted 2021-08-14; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Temporomandibular Joint Disc Displacement
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Patients diagnosed with ADD under this group are subjected to Dry Needling
  Interventions: Procedure: Dry Needling
- Test group (Experimental): Patients diagnosed with ADD under this group are administered with 1ml of PRP solution .
  Interventions: Procedure: PRP

INTERVENTIONS:
Procedure: Dry Needling — Dry Needling will be done for the patients with ADD of TMJ in the retrodiscal tissue and superior joint space .
  Arms: Control group
Procedure: PRP — Patients with ADD are administered with 1ml of PRP into the retrodiscal tissue and the superior joint space. PRP will be prepared by method proposed by Okuda et al., 2003. Reinjection will be given after 2 weeks if required.
  Arms: Test group

SUMMARY:
Pain and trismus are of the prime concerns for the patients in case of Anterior disc displacement ADD of temporomandibular joint (TMJ). In the recent times, PRP has has produced promising results in management of TMDs. It has potential healing properties on new bone and cartilage through the recruitment, proliferation, migration, and differentiation of cells and its tissue remodelling, matrix production, and chondrogenic differentiation properties. It also increases the production of hyaluronic acid by synoviocytes. Needle injury also produces immediate analgesia without hypesthesia, mainly on the painful spot making it effective for the pain reduction and improved mouth opening. Similar effect of dry needling can also be expected in the joint space where it may induce a transient inflammatory cascade leading to healing of the damaged tissue.

So, the Present study is designed to evaluate the efficacy of PRP for the treatment of ADD of TMJ.

DETAILED DESCRIPTION:
Study Design: Randomized clinical trial Study Duration: This study will be completed in 1 year 3 months (3 months for patient recruitment, 9 months for study including treatment and follow up and 3 months for data compilation).

Population: Patients suffering from Anterior Disc Displacement will be recruited in study from regular OPD of the Department of Oral Medicine and Radiology.

Sample size: Sample size consists of 39 patients in each group. Methods: PRP will be performed in test group while dry needling will be performed in control group.

ELIGIBILITY:
Inclusion Criteria:

- 1. Patients diagnosed with Anterior disc displacement clinically according to TMD/RDC criteria (2013-14).

2. Patients diagnosed with Anterior disc displacement confirmed using Magnetic Resonance Imaging.

Exclusion Criteria:

* 1. Patients with phobia to needles 2. Patients who have undergone previous treatment for anterior disc displacement in past 6 months 3. Patients with active infection at the site of injection 4. Patients on anticoagulant medication 5. Pregnancy/ Lactation 6. Patients with healing disorder or systemic disease where healing response is compromised 7. Patients with epilepsy/seizures 8. Patients with bleeding and clotting disorder 9. Patients with malignancy 10. Patients with uncontrolled para-functional habits

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2021-09-04 (Actual); Primary Completion 2023-02-15 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 2 weeks
  To evaluate the intensity of pain before and after the treatment (Visual Analogue Scale score).
Pain intensity | 4 weeks
  To evaluate the intensity of pain before and after the treatment (Visual Analogue Scale score).
Pain intensity | 3 months
  To evaluate the intensity of pain before and after the treatment (Visual Analogue Scale score).
Pain intensity | 6 months
  To evaluate the intensity of pain before and after the treatment (Visual Analogue Scale score).
Mouth opening and Functional movements | 2 weeks
  To evaluate the maximal mouth opening and functional movements before and after the treatment (millimetre).
Mouth opening and Functional movements | 4 weeks
  To evaluate the maximal mouth opening and functional movements before and after the treatment (millimetre).
Mouth opening and Functional movements | 3 months
  To evaluate the maximal mouth opening and functional movements before and after the treatment (millimetre).
Mouth opening and Functional movements | 6 months
  To evaluate the maximal mouth opening and functional movements before and after the treatment (millimetre).

SECONDARY OUTCOMES:
Joint sounds | 2 weeks
  To evaluate the changes in joint sounds before and after the treatment (present or absent ).
Joint sounds | 4 weeks
  To evaluate the changes in joint sounds before and after the treatment (present or absent ).
Joint sounds | 3 months
  To evaluate the changes in joint sounds before and after the treatment (present or absent ).
Joint sounds | 6 months
  To evaluate the changes in joint sounds before and after the treatment (present or absent ).
Pain medication | 2 weeks
  To evaluate the need for pain medicine utilization (number of tablets).
Pain medication | 4 weeks
  To evaluate the need for pain medicine utilization (number of tablets).
Pain medication | 3 months
  To evaluate the need for pain medicine utilization (number of tablets).
Pain medication | 6 months
  To evaluate the need for pain medicine utilization (number of tablets).
Patient satisfaction | 2 weeks
  To evaluate patient satisfaction before and after treatment (Likerts scale) in both groups
Patient satisfaction | 4 weeks
  To evaluate patient satisfaction before and after treatment (Likerts scale) in both groups
Patient satisfaction | 3 months
  To evaluate patient satisfaction before and after treatment (Likerts scale) in both groups
Patient satisfaction | 6 months
  To evaluate patient satisfaction before and after treatment (Likerts scale) in both groups
Sleep pattern | 2 weeks
  To evaluate sleep pattern before and after treatment (Visual Analogue Scale score) in both groups
Sleep pattern | 4 weeks
  To evaluate sleep pattern before and after treatment (Visual Analogue Scale score) in both groups
Sleep pattern | 3 months
  To evaluate sleep pattern before and after treatment (Visual Analogue Scale score) in both groups
Sleep pattern | 6 months
  To evaluate sleep pattern before and after treatment (Visual Analogue Scale score) in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No